CLINICAL TRIAL: NCT00572039
Title: Improving Function in Age-Related Macular Degeneration
Acronym: IF-AMD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Collaborators: Dartmouth College (Other); Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5U01EY015839 (NIH); NEI grant
Record Dates: First submitted 2007-12-10; First posted 2007-12-12 (Estimated); Results first posted 2015-10-15 (Estimated); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Age-Related Macular Degeneration
Keywords: Age-Related Macular Degeneration; AMD; Vision Function; Problem Solving Treatment; PST
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PST (Experimental): Problem Solving Treatment (PST)
  Interventions: Behavioral: PST
- ST (Placebo Comparator): Supportive Therapy (ST)
  Interventions: Behavioral: ST

INTERVENTIONS:
Behavioral: PST — PST will be delivered in subjects' homes over the course of 6 weeks.
  Arms: PST
Behavioral: ST — ST will be delivered in subjects' homes over the course of 6 weeks.
  Arms: ST

SUMMARY:
This randomized, controlled clinical trial will test the efficacy of Problem-Solving Treatment (PST) to improve vision function in older persons with age-related macular degeneration (AMD). AMD is a highly prevalent, disabling disease of aging that causes severe vision loss and functional decline. It is the leading cause of blindness in older persons in the United States and may affect more than 10 million people. Currently, there are no effective treatments to restore vision. Thus, improving Vision Function is a major goal of treatment. Vision function refers to vision-related abilities to perform daily living activities (e.g. reading recipes to prepare meals). Decrements in vision function will become a major public health problem as the population ages and the prevalence of AMD increases. PST is a brief, standardized, cognitive-behavioral treatment that teaches problem-solving skills.

We believe PST will enable patients with AMD find practical solutions to vision-related problems and thereby improve vision function.

We will recruit 240 AMD patients from the retina clinics of Wills Eye Institute, Philadelphia, PA, with bilateral AMD and visual acuity worse than 20/70 in the better eye. PST-trained therapists will deliver 6 1-hour, in-home sessions to the 120 subjects randomized to PST. The control treatment is Supportive Therapy (ST), a similarly structured, standardized psychological treatment that controls for the non-specific effects of treatment (n=120). ST contains no active elements beyond its non-specific components; in this way it is a placebo treatment. Independent raters, masked to treatment assignment, will assess Targeted Vision Function (primary outcome) and vision-related quality of life (secondary outcome) at 3 months to assess PST's efficacy, and at 6 months to evaluate its long-term effects. As the population ages, the disability of AMD will become more prevalent, costly, and burdensome to patients, families, and ophthalmologists. This makes devising and testing practical and affordable interventions to improve vision function a national priority.

DETAILED DESCRIPTION:
The primary hypothesis will address treatment group differences in Targeted Vision Function at 3-months, and secondary hypotheses will the long-term effect (6-months) of Problem Solving Treatment (PST) on TVF and vision-related quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Being at least 65 years old
* Having bilateral Age-Related Macular Degeneration (AMD) (atrophic or neovascular)
* Having a best corrected visual acuity of 20/70 or worse
* Moderate difficulty in at least one valued vision functional goal

Exclusion Criteria:

* Ophthalmologic Criteria. Patients who have uncontrolled glaucoma (continued visual field loss and increase in optic nerve cupping), diabetic retinopathy (due to macular edema), or cataracts for which surgery within 6 months is likely will not be eligible to participate. This information will be obtained from patients' ophthalmology charts and discussion with the patient's ophthalmologist.
* Cognitive Impairment Criteria. Cognitive functioning will be evaluated by the Project Director during the telephone screen (see Chapter 9). Patients with cognitive impairment will not be eligible to participate.
* Health Criteria. Patients with life-threatening illness (e.g., terminal cancer, need for oxygen) will not be eligible to participate. Information regarding heath status will be gleaned from patient's ophthalmology charts.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 241 (Actual)
Dates: Start 2005-08; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barry W Rovner, MD, Principal Investigator — Jefferson Medical College of Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Rovner BW, Casten RJ, Massof RW, Leiby BE, Tasman WS; Wills Eye AMD Study. Psychological and cognitive determinants of vision function in age-related macular degeneration. Arch Ophthalmol. 2011 Jul;129(7):885-90. doi: 10.1001/archophthalmol.2011.146. PMID 21746979

RESULTS

PARTICIPANT FLOW:
Groups:
- Problem Solving Treatment: Problem-solving therapy teaches problem solving skills in a structured way to enable a patient to systematically identify his or her problems, generate alternative solutions for each problem, select the best solution, develop and conduct a plan, and evaluate whether the problem is solved.
- Supportive Therapy: Supportive therapy is a structured, standardized, psychological treatment that controls for nonspecific treatment effects. Supportive therapy resembles PST in all ways but for PST's problem-solving skills training. Both interventions are based on written treatment manuals and similar in dose and intensity of attention (number and duration of sessions). Supportive therapy is nondirective and supportive, facilitates personal expression, and conveys empathy, respect, and optimism (i.e., a general sense that things can get better). The ST therapist informs subjects that ST's purpose is to explore the impact of vision loss on their lives.
Period: Overall Study
Arm/Group | Problem Solving Treatment | Supportive Therapy
Started | 121 | 120
Completed | 105 | 110
Not Completed | 16 | 10
Not completed — Withdrawal by Subject | 9 | 6
Not completed — Death | 2 | 3
Not completed — Ill | 5 | 1

BASELINE CHARACTERISTICS:
Groups:
- Problem Solving Treatment: Problem Solving Treatment (PST)
  PST: PST will be delivered in subjects' homes over the course of 6 weeks.
- Supportive Therapy: Supportive Therapy (ST)
  ST: ST will be delivered in subjects' homes over the course of 6 weeks.
- Total: Total of all reporting groups
Arm/Group | Problem Solving Treatment | Supportive Therapy | Total
Number analyzed (Participants) | 121 | 120 | 241
Age, Continuous [Mean (Standard Deviation); unit: years] | 82.7 (6.6) | 82.8 (7.3) | 82.7 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82 | 71 | 153
  Male | 39 | 49 | 88
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 120 | 119 | 239
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 121 | 120 | 241
Targeted vision function [Mean (Standard Deviation); unit: units on a scale] — At baseline subjects completed the Activities Inventory, a structured vision function questionnaire that asks patients to rate the value and difficulty of 48 vision function goal and the tasks that are required to achieve them. If a goal is important, the subject rates its "difficulty". The average TVF score is the sum of the difficulty ratings of the (up to) 4 self-selected goals divided by the number of goals (from 1 to 4). Higher average scores indicate greater disability.
  units on a scale | 2.71 (.52) | 2.73 (.52) | 2.72 (.52)
NEI VFQ-25 + supplement total score [Mean (Standard Deviation); unit: units on a scale] — We administered the 25-item National Eye Institute Vision Function Questionaire plus Supplement (NEI-VFQ).19 This version of the NEI VFQ consists of 39 items that assess self-reported vision function and vision-related QoL. The latter yields a multidimensional index of vision-related health composed of social functioning (social interactions), mental health (worry, frustration), role difficulties (accomplishing less), and dependency (relying more on others) due to vision loss. Scores range from 0 to 100, with higher scores indicating better function.
  units on a scale | 66.2 (14.3) | 65.8 (14.2) | 66.0 (14.2)
Patient Health Questionnaire-9 [Mean (Standard Deviation); unit: units on a scale] — To assess depression, we used the 9-item Patient Health Questionnaire, which yields a continuous measure of depression severity. Scores range from 0 to 27, with higher scores indicating worse depression.
  units on a scale | 1.39 (2.67) | 1.17 (2.28) | 1.28 (2.48)
Number of resources/rehabilitative devices used [Mean (Standard Deviation); unit: number of resources/devices used] | 5.14 (3.34) | 4.71 (3.02) | 4.93 (3.18)

OUTCOME MEASURES:

1. Primary Outcome: Targeted Vision Function (TVF)
Description: We identified and quantified the TVF goals that subjects valued but found difficult to achieve. To derive the TVF measure, at baseline subjects completed the Activities Inventory, a structured vision function questionnaire that asks patients to rate the value and difficulty of 48 vision function goals (e.g., daily meal preparation) and the tasks (e.g., seeing stove settings) that are required to achieve them. If a goal is important (range of 0 [not important]to 4 [very important]), the subject rates its "difficulty" (on a scale of 0 [not difficult] to 4 [impossible]). The average TVF score is the sum of the difficulty ratings of the (up to) 4 self-selected goals divided by the number of goals (from 1 to 4). Higher average scores indicate greater disability. At each outcome assessment subjects again rated the difficulty of the same targeted goals and the average TVF score was calculated.
Time Frame: 3-Months
Population: 106 PST and 112 ST participants provided data at 3 months.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Problem Solving Treatment | Supportive Therapy
Number analyzed (Participants) | 106 | 112
units on a scale | 2.18 (.88) | 2.14 (.96)
Statistical Analysis 1: Comparison: Problem Solving Treatment vs Supportive Therapy; To test the efficacy of PST to improve TVF functional reserve measures at 3 months, we used an analysis of covariance in which group differences (PST vs ST) in 3-month average TVF scores were examined, adjusting for baseline TVF score and the vision severity stratification variable. To approximate an interval scale and compensate for ceiling and floor effects, we linearized TVF scores using a logit transform. 106 PST and 112 ST participants provided data at 3 months; Test type: Superiority or Other; p = .47, ANCOVA; Mean Difference (Net) = 0.079, 95% CI 2-sided [-0.14 to 0.29]

2. Secondary Outcome: Vision-related Quality of Life
Description: We administered the 25-item National Eye Institute Vision Function Questionaire plus Supplement (NEI-VFQ).19 This version of the NEI VFQ consists of 39 items that assess self-reported vision function and vision-related QoL. The latter yields a multidimensional index of vision-related health composed of social functioning (social interactions), mental health (worry, frustration), role difficulties (accomplishing less), and dependency (relying more on others) due to vision loss. Scores range from 0 to 100, with higher scores indicating better function.
Time Frame: 3-Months
Population: 106 PST and 112 ST participants provided data at 3 months.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Problem Solving Treatment | Supportive Therapy
Number analyzed (Participants) | 106 | 112
units on a scale | 66.6 (14.9) | 65.2 (16.2)
Statistical Analysis 1: Comparison: Problem Solving Treatment vs Supportive Therapy; To test the efficacy of PST to improve NE-VFQ scores at 3 months, we used an analysis of covariance in which group differences (PST vs ST) in 3-month average NEI-VFQ scores were examined, adjusting for baseline score and the vision severity stratification variable; Test type: Superiority or Other; p = .7, ANCOVA; Mean Difference (Net) = 0.40, 95% CI 2-sided [-1.96 to 2.77]

3. Primary Outcome: Targeted Vision Function
Description: as for outcome 1
Time Frame: 6 months
Population: 105 PST and 110 ST participants provided data at 6 months.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Problem Solving Treatment | Supportive Therapy
Number analyzed (Participants) | 105 | 110
units on a scale | 2.18 (.95) | 2.15 (.96)

4. Secondary Outcome: Vision-related Quality of Life
Description: as for outcome 2
Time Frame: 6 months
Population: 105 PST and 110 ST participants provided data at 6 months.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Problem Solving Treatment | Supportive Therapy
Number analyzed (Participants) | 105 | 110
units on a scale | 66.4 (16.7) | 64.8 (17.4)

ADVERSE EVENTS:
Arm/Group | Problem Solving Treatment | Supportive Therapy
Serious Adverse Events (participants affected / at risk) | 35/121 | 29/120
Other Adverse Events (participants affected / at risk) | 0/121 | 0/120
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Problem Solving Treatment (N=121) | Supportive Therapy (N=120)
Depression (Psychiatric disorders) | 5 (5) | 1 (1)
Fall (Musculoskeletal and connective tissue disorders) | 6 (6) | 8 (8)
Amputation (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Congestive Heart Failure (Cardiac disorders) | 2 (2) | 3 (3)
Death due to CHF (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac event (Cardiac disorders) | 4 (4) | 2 (2)
Stroke (Vascular disorders) | 3 (3) | 2 (2)
Dehydration/anemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Knee pain/back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (5)
hypoglycemia (Endocrine disorders) | 1 (1) | 0 (0)
Varicosities (Vascular disorders) | 1 (1) | 0 (0)
Death NOS (General disorders) | 2 (2) | 1 (1)
Pagets diesease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Subdural hematoma (Vascular disorders) | 0 (0) | 1 (1)
Fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Severe reflux, Hiatal hernia, Bowel obstruction (Gastrointestinal disorders) | 3 (3) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Myasthenia Gravis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No